CLINICAL TRIAL: NCT01630746
Title: A Randomized, Double-Blind, Multicenter Study to Evaluate the Acid-inhibitory and Dose-response Efficacy of TAK-438 (20 mg, 40 mg) in Patients With Proton Pump Inhibitor (PPI) - Resistant Erosive Esophagitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: TAK-438/OCT-002; JapicCTI-121882 (Registry Identifier: JapicCTI); U1111-1130-9074 (Registry Identifier: WHO)
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-02

CONDITIONS: Erosive Esophagitis
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

ARMS (2):
- TAK-438 20 mg/day (Experimental)
  Interventions: Drug: TAK-438
- TAK-438 40 mg/day (Experimental)
  Interventions: Drug: TAK-438

INTERVENTIONS:
Drug: TAK-438
  Arms: TAK-438 20 mg/day
Drug: TAK-438
  Arms: TAK-438 40 mg/day

SUMMARY:
The purpose of this study is to evaluate the acid-inhibitory and dose-response efficacy of TAK-438 (20 mg, 40 mg) in patients with PPI-resistant erosive esophagitis.

ELIGIBILITY:
Inclusion Criteria:

1. The participant has been treated with standard-dose or higher-than-standard-dose PPI until immediately before the start of the Observation Phase.
2. Outpatient (in principle)
3. At the endoscopy scheduled for the Observation Phase (Visit 2), the participant must have endoscopically confirmed reflux esophagitis of Grade A to D, as defined by the LA classification grading system, which remains insufficiently controlled with standard-dose or higher-than-standard-dose PPI therapy.
4. The participant showed good compliance to the study medication in the Observation Phase (compliance rate 80% or more).

Exclusion Criteria:

1. Participants with an esophagus-related complication (eosinophilic esophagitis, esophageal varices, scleroderma, viral or fungal infection, esophageal stenosis, etc.), a history of radiotherapy or cryotherapy of the esophagus, a caustic or physiochemical trauma (esophageal sclerotherapy, etc.). However, participants with Schatzki's ring (mucosal tissue ring around inferior esophageal sphincter) or Barrett's esophagus are allowed to be included.
2. Participants who have received surgery or treatment affecting gastroesophageal reflux (cardioplasty, dilation of esophageal stenosis [excluding Schatzki's ring], etc.), or who have a history of surgery of stomach or duodenum (excluding removal of benign polyp under endoscopy)
3. Participants who have acute upper gastrointestinal bleeding, gastric or duodenal ulcer (mucosal defect with white coating) at the start of the Observation Phase (Visit 1) or at endoscopy during the Observation Phase (Visit 2) . However, participants with gastric or duodenal erosions are allowed to be included.
4. Participants with a previous or current history of Zollinger-Ellison syndrome, or other gastric acid hypersecretion disorders.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Time-course of changes in 24-hour gastroesophageal pH | Week 8
  Gastric and esophageal pH4 HTR (pH 4 Holding Time Ratio) will be calculated based on 24-hour gastroesophageal pH monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (11):
- Japan (11):
  - Gifu, Gifu
  - Sapporo, Hokkaido
  - Hitachi-shi, Ibaraki
  - Kochi, Kochi
  - Sendai, Miyagi
  - Osaka, Osaka
  - Saga, Saga-ken
  - Izumo-shi, Shimane
  - Hamamatsu, Shizuoka
  - Bunkyo-ku, Tokyo
  - Mitaka-shi, Tokyo